CLINICAL TRIAL: NCT02421354
Title: Phase 2 Study of Nivolumab in Patients With Primary Myelofibrosis, Post-Essential Thrombocythemia Myelofibrosis, or Post-Polycythemia Vera Myelofibrosis
Brief Title: Nivolumab in Treating Patients With Primary Myelofibrosis, Post-Essential Thrombocythemia Myelofibrosis, or Post-Polycythemia Vera Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0962; NCI-2015-00836 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0962 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-04-10; First posted 2015-04-20 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Hepatomegaly; Myelofibrosis Transformation in Essential Thrombocythemia; Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Primary Myelofibrosis; Splenomegaly
MeSH Terms: conditions — Hepatomegaly; Polycythemia Vera; Primary Myelofibrosis; Splenomegaly | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 60 minutes once every 2 weeks for 8 doses and then once every 12 weeks thereafter. Treatment may continue for up to 4 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well nivolumab works in treating patients with primary myelofibrosis, post-essential thrombocythemia myelofibrosis, or post-polycythemia vera myelofibrosis. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy/clinical activity of nivolumab in patients with myelofibrosis (MF).

SECONDARY OBJECTIVES:

I. To determine the safety of nivolumab in patients with MF.

TERTIARY OBJECTIVES:

I. To explore time to response and duration of response. II. To assess changes in symptom burden. III. To explore changes in bone marrow fibrosis. IV. To explore changes in Janus kinase 2 valine at amino acid position 617 (JAK2V617F) (or other molecular marker) allele burden or changes in cytogenetic abnormalities.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 60 minutes once every 2 weeks for 8 doses and then once every 12 weeks thereafter. Treatment may continue for up to 4 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30, 60, and 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MF (either primary or post essential thrombocythemia/polycythemia vera) requiring therapy, including those previously treated and relapsed or refractory, or if newly diagnosed, with intermediate-1 or -2 or high risk according to International Prognostic Scoring System (IPSS)
* Previously treated with ruxolitinib (unless not a good candidate for ruxolitinib therapy in the judgment of treating physician)
* Palpable splenomegaly or hepatomegaly of more than or equal to 5 cm below left or right, respectively, costal margin on physical exam
* Understanding and voluntary signing an institutional review board (IRB)-approved informed consent form
* No prior history of immune checkpoint modulator therapy
* Disease-free of other malignancies
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Negative pregnancy test in females of childbearing potential (FCBP); male patients with female partners of child-bearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 23 weeks (for females) or 31 weeks (for males) following the last dose of study medication; acceptable forms of contraception include 1 highly effective method such as an intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation, or partner's vasectomy and at least 1 additional approved barrier method such as a latex condom, diaphragm, or cervical cap plus spermicide; female patients of childbearing potential must not be breast-feeding or planning to breast feed and must have a negative pregnancy test within 24 hours of the first study treatment
* Direct bilirubin equal to or less than 1.5 x upper limit of normal (ULN)
* Serum creatinine equal to or less than 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) equal to or less than 2.5 x ULN (unless considered to be related to MF or patient has known history of Gilberts, in which case it must be equal to or less than 5 x ULN)

Exclusion Criteria:

* Use of any other standard or experimental therapy within 14 days of starting study therapy
* Lack of recovery from all toxicity from previous therapy to grade 1 or baseline
* Any concurrent severe and/or uncontrolled medical conditions that could increase the patient's risk for toxicity while in the study or that could confound discrimination between disease- and study treatment-related toxicities
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association class III-IV within 6 months prior to their first dose of the study drugs
* Patients who are currently receiving chronic (> 14 days) treatment with corticosteroids at a dose equal to or more than 10 mg of prednisone (or its glucocorticoid equivalent) per day, or any other chronic immunosuppressive treatment that cannot be discontinued prior to starting study drug
* Patients with autoimmune diseases are excluded: patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis)
* Pregnant or breast feeding (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive beta-human chorionic gonadotropin (HCG) laboratory test
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C
* The use of dietary supplements or herbal medications within 7 days of starting study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2015 to October 2017
Period: Overall Study
Arm/Group | Treatment (Nivolumab)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 74 [69 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate, Defined as Complete Remission + Partial Remission + Clinical Improvement
Description: Responses will be categorized according to the revised International Working Group-Myeloproliferative Neoplasms Research and Treatment and European LeukmiaNet consensus criteria for myelofibrosis.
Time Frame: 14 weeks (after 8 doses of therapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 3/8
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=8)
Abdominal Pain (General disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Back Pain (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Esophageal Varices Hemorrhage (Gastrointestinal disorders) | 1 (1)
Facial Nerve Disorder (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Fever (General disorders) | 1 (2)
Gastric Hemorrhage (Gastrointestinal disorders) | 2 (4)
Headache (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=8)
Pain (General disorders) | 3 (5)
Neutropenic Fever (Infections and infestations) | 1 (1)
Leptomeningeal disease (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Infection (Infections and infestations) | 3 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 1 (1)
Increased Transaminases (Investigations) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Cardiomegaly (Cardiac disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Edema (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Elevated Alkaline Phophatase (Investigations) | 1 (1)
Elevated Creatinine (Investigations) | 1 (1)
Esophageal Varicies (Gastrointestinal disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemotympanum (Ear and labyrinth disorders) | 1 (1)
Hepatobiliary disorder (Hepatobiliary disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Hemorrhage (Nervous system disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Renal lesion (Renal and urinary disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT02421354/Prot_SAP_000.pdf